CLINICAL TRIAL: NCT01721330
Title: A Double-Blind Comparison of Naltrexone and Placebo in Adults With Attention Deficit Hyperactivity Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Competing studies
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P-002252
Record Dates: First submitted 2012-10-30; First posted 2012-11-05 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Psychopharmacology; Psychiatry; Non-stimulant treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Active Comparator): Active Naltrexone administered twice daily up to a maximum total dose of 100mg/day.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Naltrexone-masked placebo administered twice daily up to a maximum total dose of 100mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Up to 100mg of Naltrexone once a day for 6 weeks
  Arms: Naltrexone
Drug: Placebo — Placebo twice a day for 6 weeks
  Arms: Placebo

SUMMARY:
The primary aim of this study is to assess whether naltrexone as a monotherapy is effective in treating ADHD in adults. Medications that increase dopamine are often effective treatments for ADHD. Since naltrexone is a kappa opioid receptor antagonist, it increases dopamine in the brain. The investigators predict that naltrexone as a monotherapy will be effective for ADHD symptoms in adults with ADHD.

The investigators also plan to assess the effects of naltrexone on dopamine as measured by changes in serum prolactin. The investigators predict that naltrexone will increase dopamine as indexed by decreases in serum prolactin. This study will be a six-week, double-blind, placebo-controlled pilot study with adults 18-55 years of age with ADHD.

DETAILED DESCRIPTION:
This will be a six-week, randomized, double-blind, placebo-controlled, parallel design study of adult ADHD with naltrexone monotherapy. Eligible and consenting subjects will be recruited into the study. The first visit will consist of a meeting with a study clinician who obtains consent, assesses for eligibility, and completes study rating scales. After this evaluation, subjects will complete a neuropsychological assessment and study rating scales (two hours; this visit can take place over multiple days, if necessary). Subjects will then be randomized to naltrexone (50 mg) once a day with breakfast or placebo at a ratio of 1:1 to be increased, if tolerated, to 100 mg by week 1.

Blood will be drawn for prolactin, basic metabolic panel, CBC, and LFT's at pre-baseline and upon completion of the study. Ten cc's (approximately two teaspoons) of blood will be required for the basic metabolic panel, CBC, and LFT's at each drawing. An additional five cc's (approximately one teaspoon) of blood will be required for laboratory testing of prolactin levels at each drawing. Dipstick urine drug testing will be done at pre-baseline.

Women of child bearing age will also have a urine pregnancy test at pre-baseline.

Although every effort will be made to encourage subjects to keep regularly scheduled appointments, in the event that a subject is unable to come into the office within a reasonable timeframe of a scheduled visit, and the treating research clinician feels that subject safety will not be jeopardized by doing so, the clinician can conduct the visit with the subject over the telephone. However, study evaluation visit (pre-baseline), baseline visit, mid-point visit (week 3), or the final study visit may not be conducted over the phone. Additionally, phone visits may not occur for two consecutive visits.

ELIGIBILITY:
Inclusion Criteria

1. Male and female outpatients 18-55 years of age.
2. Diagnosis of ADHD, by Diagnostic and Statistical Manual-IV (DSM-IV) by clinical evaluation by an expert clinician.
3. A CGI of 7 (among the most extremely ill patients) at the pre-baseline visit is exclusionary, and any subject who presents a CGI-S of 7 at any point during the study will be removed from participation.
4. Subjects presenting with a CGI-S score of 6 (severely ill) at two consecutive visits after week 2 will be dropped from the study (i.e. A subject with a CGI of 6 at his/her week 3 visit and at week 4 visit will be dropped from the study at the week 4 visit). Subjects who are dropped for severe or worsening symptoms after exposure to the study medication will receive free follow up care as described in the detailed protocol and protocol summary.
5. Subjects treated for anxiety disorders and depression who are on a stable medication regimen for at least one month, and who have a disorder-specific CGI-Severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-Anxiety rating scales below 15 (mild range).

Exclusion Criteria

1. Any clinically unstable psychiatric conditions including any history of psychosis or mania, suicidality, sociopathy, criminality, or delinquency.
2. Current (last 3 months) substance use disorders (alcohol or drugs),
3. Medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study including cardiovascular disease, current untreated hypertension, or history of renal or hepatic impairment.
4. A condition that will or may require treatment with opioid analgesics.
5. Clinically significant abnormal baseline laboratory LFT's, which is defined as LFT's greater than the ULN.
6. Mental retardation (IQ < 80).
7. Organic brain disorders including delirium, dementia, seizures, stroke, neurosurgery, and head trauma with loss of consciousness.
8. Pregnant or nursing females.
9. Subjects with current adequate treatment for ADHD.
10. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol (a stable and effective treatment regimen of an SSRI or benzodiazepine is permitted per clinical review).
11. Non-English speaking subjects will not be allowed into the study for the following reasons:

    1. The assessment instruments are unavailable and have not been adequately standardized in other languages;
    2. Even if such translation services were available, the assessments in the English language conducted by English-speaking clinicians and raters with English-speaking subjects are already extremely time-consuming, lasting many hours, making it unfeasible, unrealistic, and of dubious clinical validity to conduct them with a translator with non-English-speaking subjects;
    3. Psychiatric questionnaires and evaluations are taxing, and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.33 (NA) — Only one subject | 32.21 (2.13) | 33.58 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult Investigator Symptom Rating Scale (AISRS) Score
Description: The AISRS is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (none) to 3 (severe). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). We measured the change in AISRS score from baseline to week 6.
Time Frame: 6 weeks
Population: One subject withdrew from the study before receiving study medication, so data from only two subjects was analyzed (one subject in each group). Therefore, means and standard deviations were not calculated.
Measure: Number; unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | -6.0 | -5.0

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=1) | Placebo (N=2)
Flu (General disorders) | 1 (1) | 0 (0)
Muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prior to completion due to competing studies. Therefore, only one subject in each group was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes